CLINICAL TRIAL: NCT06327737
Title: Contribution of End-Tidal Carbon Dioxide and Integrated Pulmonary Index Monitoring With Capnography to Diabetic Ketoacidosis Diagnosis and Management
Brief Title: Diabetic Ketoacidosis Diagnosis and Management
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Collaborators: Ceren Kahraman (Unknown)
Responsible Party: Principal Investigator, Ozlem Tolu Kendir, Assoc. Prof., Akdeniz University
Other Study IDs: AKDENIZ-KAEK-916
Record Dates: First submitted 2024-03-06; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Metabolic Acidosis; Diabetic Ketoacidosis; Brain Edema
Keywords: Type 1 diabetes mellitus (Type 1 DM); Diabetic Ketoacidosis (DKA); Capnography; Blood gas; Integrated Pulmonary Index; End tidal Carbon Dioxide (EtCO2)
MeSH Terms: conditions — Acidosis; Diabetic Ketoacidosis; Brain Edema; Diabetes Mellitus, Type 1 | interventions — Capnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Capnography — This is non-invasive follow-up method to the management of DKA and the reduction of the frequency of invasive procedures was investigated in patients diagnosed with diabetic ketoacidosis (DKA) in the pediatric emergency department and followed up with capnography.

SUMMARY:
This is the first and only study conducted on the use of capnography in children diagnosed with DKA to evaluate the initial clinical grading of DKA, monitor clinical improvement, and predict complications such as brain edema.

DETAILED DESCRIPTION:
Purpose: In this study, the contribution of this non-invasive follow-up method to the management of DKA and the reduction of the frequency of invasive procedures was investigated in patients diagnosed with diabetic ketoacidosis (DKA) in the pediatric emergency department and followed up with capnography

Method: This study is a prospective clinical study. Between October 2020- November 2022, EtCO2 and IPI follow-up of 0-18 year-old pediatric patients diagnosed with DKA in the Pediatric Emergency Service of Akdeniz University Medical Faculty Hospital was performed by capnography. DKA diagnosis, grading, clinical follow-up and treatment termination criteria of the patients were determined according to the ISPAD 2018 Diagnosis and Treatment Guidelines. In the study; During the clinical follow-up, changes in GCS, blood glucose, vital, blood gas and capnograph parameters were examined. Demographic data were analyzed in all patients and in groups of patients who underwent DKA grading. GCS, blood gas and capnograph parameters were compared in the patient groups with DKA grading. Diagnostic test performances of blood gas and capnograph parameters were compared to detect low GCS

ELIGIBILITY:
Inclusion Criteria:

* The study group consisted of pediatric patients aged 0-18 years who were diagnosed with Diabetic Ketoacidosis and applied to Akdeniz University pediatric emergency department.
* Written consent was obtained.

Exclusion Criteria:

• Who did not give written consent were not included in the study.

Ages: 15 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: During the study, 55 of 66 patients diagnosed with DKA in the pediatric emergency department of our hospital were included in the study. One of our patients was during the researcher's leave; 7 of them were excluded from the study because they were in periods when capnograph cannula was not available in our hospital and 3 of them were excluded due to patient non-compliance.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Correlation between PCO2 and EtCO2 | 2 days
  The positive linear correlation between PCO2 and EtCO2 indicates that acidosis can be monitored with EtCO2.
Correlation between Integrated Pulmonary Index and degree of acidosis | 2 days
  Detection of a positive linear correlation between those with Integrated Pulmonary Index <8 and the degree of acidosis
Prediction of cerebral edema with Integrated Pulmonary Index | 2 days
  Detection of significant decrease in Glasgow Coma Scale (GCS<13) in patients with Integrated Pulmonary Index <4

CONTACTS AND LOCATIONS:
Overall Officials: OZLEM TOLU KENDIR, Assoc. Prof., Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

REFERENCES:
- [Derived] Kendir OT, Kahraman C, Tekerek NU, Gurlu R, Parlak M, Erkek N. The contribution of end-tidal carbon dioxide monitoring to the management of pediatric patients with diabetic ketoacidosis. Am J Emerg Med. 2026 Jan;99:151-154. doi: 10.1016/j.ajem.2025.09.050. Epub 2025 Sep 26. PMID 41033061